CLINICAL TRIAL: NCT06168019
Title: Influenza & COVID-19 Obstetric and Perinatal Epidemiology (ICOPE) Study in India
Brief Title: Influenza & COVID-19 Obstetric and Perinatal Epidemiology Study in India
Acronym: ICOPE
Status: Recruiting | Type: Observational
Sponsor: Boston University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Lata Medical Research Foundation, Nagpur (Other)
Responsible Party: Sponsor
Other Study IDs: H-43541; UG1HD078439 (NIH)
Record Dates: First submitted 2023-12-12; First posted 2023-12-13 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Influenza; COVID-19; SARS-COV-2 Infection; Other Respiratory Viruses; Perinatal Morbidity; Infant Morbidity
Keywords: Pregnant women; Government Medical College Hospital, Nagpur, India; Covid-19 vaccination; Antenatal care; Postpartum
MeSH Terms: conditions — Influenza, Human; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for COVID-19, influenza and ORV antibodies and potential modifiers of infection will be drawn at a maximum of four time points - baseline (week 6-13 of pregnancy), at study visit 3 (week 28-34), at study visit 4 (week 37-prior to delivery) of pregnancy and between delivery and day 42-70 postpartum/after miscarriage. In addition a random subset of 200 subjects will be invited to provide nasopharyngeal (NP)swabs during all 4 study visits and between delivery and day 7 postpartum (prior to discharge) to track asymptomatic viral infection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Influenza & COVID-19 Obstetric and Perinatal Epidemiology (ICOPE): Pregnant women in their first trimester of pregnancy who present to the outpatient antenatal care clinic at Government Medical College Hospital in Nagpur, India.
  Interventions: Other: Exposures

INTERVENTIONS:
Other: Exposures — COVID-19, Influenza and ORV impact on the pregnant woman, her fetus and newborn

SUMMARY:
This study will be conducted as a prospective cohort study, enrolling all eligible women in their first trimester of pregnancy during a baseline visit during week 6-13 of pregnancy at Government Medical College Hospital, Nagpur. The Hospital provides primary, secondary, and tertiary care and the obstetric department delivers about 10,000 babies a year. The hypothesis is that co-infection of other respiratory viruses (ORV), particularly COVID-19 and Influenza increases the risk of adverse pregnancy outcomes in mothers and babies and could address the current standard of care in India to not vaccinate pregnant women during pregnancy, by either encouraging vaccination against both viruses before planning a pregnancy or during pregnancy based on global data supporting the safety of this strategy.

DETAILED DESCRIPTION:
All pregnant women enrolled in the study will receive standard of care throughout their pregnancy, labor and delivery and post-partum to discharge. Wherever possible, study visits will coincide with regular antenatal (ANC) care and blood draws will be added to standard blood draws during ANC, labor and delivery and postpartum care. Women will be counselled about procedure to reduce the risk of acquiring ORV during pregnancy. Since this study is observational, we do not anticipate any specific safety concerns with study interviews and procedures, but the investigators will monitor potential adverse events to determine if they are likely or possibly study related.

PRIMARY OBJECTIVE: Determine the prevalence, incidence, and maximal severity of symptomatic or asymptomatic COVID-19 in pregnant women to day 42 postpartum/after miscarriage on maternal outcomes. Secondary analysis will evaluate whether influenza/Other Respiratory Viruses (ORV) infection or COVID-19 vaccination modifies or mediates this risk.

SECONDARY OBJECTIVE: Determine the effect of maternal COVID-19 infection on the fetus and/or neonate during pregnancy through day 7 of life. Secondary analysis will focus on whether influenza/ORV or vaccination modifies, and pre-term birth mediates this risk.

EXPLORATORY OBJECTIVE: Characterize patterns and trajectories of host response/ inflammatory biomarkers as potential mediators of COVID-19 ± Influenza and ORV infection on progression to severe illness in pregnant women/mothers admitted to Government Medical College hospital with COVID-19. Modifiers include COVID-19 , Influenza and other ORV vaccinations.

ELIGIBILITY:
Inclusion Criteria:

Women aged 18 to 50 years registering for antenatal care (ANC) at Government Medical College Hospital (GMC) Nagpur, India

* Estimated Gestational Age at registration <14 weeks based on ultrasound report at the baseline study visit;
* Intends to receive pregnancy, labor and delivery and neonatal care at GMC;
* Plans to live within the city limits of Nagpur throughout their pregnancy and labor and delivery to facilitate access to GMC for evaluation of ILI and COVID-19 symptoms;
* Willing to be contacted two times per week by call or text for ILI/ COVID-19 symptom screening and return to GMC for evaluation and an NP swab/evaluation if symptoms are reported;
* Willing to take temperature with the provided digital thermometer, and maintain a symptom diary after training;
* Willing to provide information on pregnancy and neonatal outcomes if care occurs outside GMC;
* Willing to permit venous blood draws on at least 4 timepoints --1) Baseline study visit, 2)28-34 weeks, 3) 37 weeks - prior to delivery and 4) after delivery;
* Willing to permit blood draws if hospitalized at GMC for COVID-19 infection;
* Willing to consent to participate in the study

Exclusion Criteria:

* Anyone who is deemed to have limited decision-making capacity as defined by Boston University IRB i.e. Substantial impairment of cognitive functions (e.g. attention, comprehension, memory, and intellect), or conditions that might affect their cognitive functions.
* Anyone who is deemed to have limited capacity to consent as defined by Boston University Institutional Review Board (IRB) i.e. The ability to provide legally effective consent to enroll in a research study (AAHRPP definition).

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: The study population is pregnant women in their first trimester of pregnancy who present to the outpatient antenatal care clinic at Government Medical College Hospital in Nagpur, India. Women will be aged 18-50 and can be from any race or ethnic group.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-12-26 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Maternal composite adverse outcome variable | 1 year
  The maternal composite variable includes any of following 3 outcomes:
  * Preterm labour, defined as hospitalization for the management of onset of labor before fetus age 37 weeks, regardless of when birth occurs;
  * Pre-eclampsia with severe features, defined as the new onset of systolic blood pressure >160 mm Hg and/or diastolic blood pressure >110 mm Hg and proteinuria (World Health Organization (WHO) definition);
  * Mortality at any time between enrolment and day 42 post-partum/after miscarriage.

SECONDARY OUTCOMES:
Perinatal composite adverse outcome variable | 1 year
  The perinatal adverse outcomes includes any of the following 3 outcomes:
  * Preterm birth, defined as gestational age of <37 weeks at birth, based on gestational age dating by ultrasound obtained before study enrolment;
  * Neonatal critical illness, defined as any sign of critical illness in the newborn and/or continued hospitalization after day 7 of life;
  * Perinatal Mortality, defined as fetal mortality after week 20 of pregnancy through neonatal death by day 7 of life

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Hibberd, MD PhD, Principal Investigator — Boston University School of Public Health, Global Health; Archana Patel, MD, Principal Investigator — Lata Medical Research Foundation, Nagpur India
Locations (2):
- Boston University School of Public Health, Global Health, Boston, Massachusetts, United States
- Government. Medical College Hospital, Nagpur, India

IPD SHARING:
Plan to Share IPD: Undecided